CLINICAL TRIAL: NCT01945775
Title: A PHASE 3, OPEN-LABEL, RANDOMIZED PARALLEL,2-ARM,MULTI-CENTER STUDY OF TALAZOPARIB(BMN 673) VERSUS PHYSICIAN'S CHOICE IN GERMLINE BRCA MUTATION SUBJECTS WITH LOCALLY ADVANCED AND/OR METASTATIC BREAST CANCER, WHO HAVE RECEIVED PRIOR CHEMOTHERAPY REGIMENS FOR METASTATIC DISEASE
Brief Title: A Study Evaluating Talazoparib (BMN 673), a PARP Inhibitor, in Advanced and/or Metastatic Breast Cancer Patients With BRCA Mutation (EMBRACA Study)
Acronym: EMBRACA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 673-301; C3441009 (Other: Alias Study Number); 2013-002716-28 (EudraCT Number); U1111-1155-7579 (Other: Universal Trial Number)
Record Dates: First submitted 2013-09-11; First posted 2013-09-19 (Estimated); Results first posted 2018-10-03 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2021-12

CONDITIONS: Breast Neoplasms; BRCA 1 Gene Mutation; BRCA 2 Gene Mutation
Keywords: Breast cancer; BRCA mutation; PARP inhibitor; BRCA 1; BRCA 2
MeSH Terms: conditions — Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- talazoparib (Experimental): Patient will be randomized 2:1 to receive talazoparib oral capsules (1.0 mg) once daily for 21 continuous days
  Interventions: Drug: talazoparib
- Physician's-Choice (Active Comparator): Capecitabine, Eribulin, Gemcitabine or Vinorelbine
  Interventions: Drug: Physician's-Choice

INTERVENTIONS:
Drug: talazoparib — Until progression or unacceptable toxicity develops
  Arms: talazoparib
Drug: Physician's-Choice — Capecitabine, Eribulin, Gemcitabine or Vinorelbine
  Arms: Physician's-Choice

SUMMARY:
The purpose of this open-label, 2:1 randomized phase III trial is to compare the safety and efficacy of talazoparib (also known as BMN 673) versus protocol-specific physician's choice in patients who have locally advanced and/or metastatic breast cancer with germline BRCA mutations.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma of the breast
* Locally advanced breast cancer that is not amenable to curative radiation or surgical cure and/or metastatic disease appropriate for systemic single cytotoxic chemotherapy
* Documentation of a deleterious, suspected deleterious, or pathogenic germline BRCA1 or BRCA2 mutation from Myriad Genetics or other laboratory approved by the Sponsor
* No more than 3 prior chemotherapy-inclusive regimens for locally advanced and/or metastatic disease (no limit on prior hormonal therapies or targeted anticancer therapies such as mechanistic target of rapamycin (mTOR) or CDK4/6 inhibitors, immune-oncology agents, tyrosine kinase inhibitors, or monoclonal antibodies against CTL4 or VEGF)
* Prior treatment with a taxane and/or anthracycline in the neoadjuvant, adjuvant, locally advanced, or metastatic setting unless medically contraindicated
* Have measurable or non-measurable, evaluable disease by the revised response evaluation criteria in solid tumors (RECIST) v.1.1
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* First-line locally advanced and/or metastatic breast cancer with no prior adjuvant chemotherapy unless the Investigator determines that one of the 4 cytotoxic chemotherapy agents in the control arm would otherwise be offered to the subject
* Prior treatment with a PARP inhibitor (not including iniparib)
* Not a candidate for treatment with at least 1 of the treatments of protocol-specific physician's choice (ie, capecitabine, eribulin, gemcitabine, vinorelbine)
* Subjects who had objective disease progression while receiving platinum chemotherapy administered for locally advanced or metastatic disease; subjects who received low-dose platinum therapy administered in combination with radiation therapy are not excluded
* Subjects who have received platinum in the adjuvant or neoadjuvant setting are eligible; however, subjects may not have relapsed within 6 months of the last dose of prior platinum therapy
* Cytotoxic chemotherapy within 14 days before randomization
* Radiation or anti-hormonal therapy or other targeted anticancer therapy within 14 days before randomization
* HER2 positive breast cancer
* Active inflammatory breast cancer
* CNS metastases

  * Exception: Adequately treated brain metastases documented by baseline CT or MRI scan that has not progressed since previous scans and that does not require corticosteroids (except prednisone ≤ 5 mg/day or equivalent) for management of CNS symptoms. A repeat CT or MRI following the identification of CNS metastases (obtained at least 2 weeks after definitive therapy) must document adequately treated brain metastases.
  * Subjects with leptomeningeal carcinomatosis are not permitted
* Prior malignancy except for any of the following:

  * Prior BRCA-associated cancer as long as there is no current evidence of the cancer
  * Carcinoma in situ or non-melanoma skin cancer
  * A cancer diagnosed and definitively treated ≥ 5 years before randomization with no subsequent evidence of recurrence
* Known to be human immunodeficiency virus positive
* Known active hepatitis C virus, or known active hepatitis B virus
* Known hypersensitivity to any of the components of talazoparib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2021-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (346):
- United States (193):
  - Arizona Oncology Associates P.C. - NAHOA, Flagstaff, Arizona
  - HonorHealth, Scottsdale, Arizona
  - Virginia G. Piper Cancer Pharmacy, Scottsdale, Arizona
  - Kaiser Permanente Medical Center Lab Drawing Station, Antioch, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Fairfield, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Gilroy, California
  - Los Angeles Hematology Oncology Medical Group, Glendale, California
  - Marin Specialty Care, Greenbrae, California
  - Los Angeles Hematology Oncolgy Medical Group, Los Angeles, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Drug Management Only: UCLA West Medical Pharmacy, Attn:Steven L. Wong, Pharm.D., Los Angeles, California
  - Drug Management only: UCLA West Medical Pharmacy, Los Angeles, California
  - UCLA West Medical Pharmacy, Attn: Steven L. Wong, Pharm. D., Los Angeles, California
  - UCLA West Medical Pharmacy, Attn: Steven L. Wong, Pharm.D., Los Angeles, California
  - UCLA West Medical Pharmacy, Attn: Steven L. Wong, Los Angeles, California
  - UCLA West Medical Pharmacy, Attn:Steven L. Wong, Pharm.D., Los Angeles, California
  - Regulatory Managment Only: TRIO-US Central Administration, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - TRIO-US Central Administration, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Martinez, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Milpitas, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Modesto, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Mountain View, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Napa, California
  - Kaiser Permanente Medical Center (clinic+DSL), Oakland, California
  - Kaiser Permanente Medical Center (Radiology), Oakland, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Pleasanton, California
  - Torrance Health Association, DBA Torrance Memorial Physician Network/Cancer care Associates, Redondo Beach, California
  - Kaiser Permanente Medical Center Lab Drawing Station, Redwood City, California
  - Kaiser Permanente Medical Center (clinic+DSL), Roseville, California
  - Southern California Permanente Medical Group, San Diego, California
  - UCSF - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - UCSF Helen Diller Comprehensive Cancer Centre - Precision Cancer Medicine Building, San Francisco, California
  - Kaiser Permanente Mission Bay Medical Center Lab Drawing Station, San Francisco, California
  - Kaiser Permanente Medical Center Lab Drawing Station, San Jose, California
  - Kaiser Permanente Medical Center (clinic+DSL), San Leandro, California
  - Pacific Central Coast Health Centers - San Luis Obispo Oncology and Hematology Health Center, San Luis Obispo, California
  - Ridley Tree Cancer Center, Santa Barbara, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Kaiser Permanente Medical Center (clinic+DSL), Santa Clara, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - UCLA Hematology Oncology, Santa Monica, California
  - UCLA Hematology/Oncology - Parkside, Santa Monica, California
  - UCLA Santa Monica Medical Center & Orthopaedic Hospital, Santa Monica, California
  - Sutter North Bay Health Plaza, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Sutter Santa Rosa Regional Hospital, Santa Rosa, California
  - Ridley Tree Cancer Center, Solvang, California
  - Kaiser Permanente Medical Center (clinic+DSL), South San Francisco, California
  - Stanford Cancer Institute, Stanford, California
  - Stanford Women's Cancer Center, Stanford, California
  - UCLA Hematology/Oncology - Santa Clarita, Valencia, California
  - Kaiser Permanente Medical Center (clinic+DSL), Vallejo, California
  - Kaiser Permanente Medical Center (clinic+DSL), Walnut Creek, California
  - Southern California Permanente Medical Group, Woodland Hills, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Rocky Mountain Cancer Centers, Boulder, Colorado
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, Littleton, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Longmont, Colorado
  - Rocky Mountain Cancer Centers, Parker, Colorado
  - Rocky Mountain Cancer Centers, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, Thornton, Colorado
  - Cancer Center of Central Connecticut, Plainville, Connecticut
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Sylvester Comprehensive Cancer Center Deerfield Beach, Deerfield Beach, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Florida Cancer Specialists, Hudson, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville Beach, Florida
  - Florida Cancer Specialists, Lady Lake, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Lecanto, Florida
  - "University of Miami Hospital & Clinics,Sylvester Comprehensive Cancer Center/UMHC", Miami, Florida
  - Sylvester Comprehensive Cancer Center Kendall, Miami, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Orlando Health, Inc, Orlando, Florida
  - Sylvester Comprehensive Cancer Center Plantation, Plantation, Florida
  - Cancer Specialists of North Florida, Saint Augustine, Florida
  - Florida Cancer Specialists, Spring Hill, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Central Georgia Cancer Care, PC, Macon, Georgia
  - Central Georgia Cancer Care, PC, Warner Robins, Georgia
  - Indiana University- Melvin and Bren Simon Cancer Center (IUSCC), Indianapolis, Indiana
  - IU Health University Hospital, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Clinic, Indianapolis, Indiana
  - The University of Kansas Cancer Center (Regulatory Office), Fairway, Kansas
  - The University of Kansas Cancer Center, Kansas City, Kansas
  - The University of Kansas Cancer Center, Overland Park, Kansas
  - The University of Kansas Cancer Center - Investigational Drug Services, Westwood, Kansas
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - University of Michigan Health System, Ann Arbor, Michigan
  - Cancer And Hematology Centers Of Western Michigan, Grand Rapids, Michigan
  - Minnesota Oncology Hematology, P.A., Coon Rapids, Minnesota
  - Minnesota Oncology Hematology, P.A., Edina, Minnesota
  - Minnesota Oncology Hematology, P.A., Fridley, Minnesota
  - Minnesota Oncology Hematology, P.A., Maplewood, Minnesota
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Minnesota Oncology Hematology, P.A., Saint Paul, Minnesota
  - Minnesota Oncology Hematology, P.A., Woodbury, Minnesota
  - The West Clinic, P.C., Corinth, Mississippi
  - The West Clinic, P.C. d/b/a West Cancer Center, Southaven, Mississippi
  - The University of Kansas Cancer Center, Kansas City, Missouri
  - The University of Kansas Cancer Center, Lee's Summit, Missouri
  - Comprehensive Cancer Centers Of Nevada, Henderson, Nevada
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Oncology Hematology, P.C., Clifton Park, New York
  - New York University Langone Medical Center, New York, New York
  - Perlmutter Cancer Center, New York, New York
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Weill Cornell Breast Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - Eastchester Center for Cancer Care, The Bronx, New York
  - Hope Women's Cancer Centers, Asheville, North Carolina
  - MH Mission Hospital, LLLP, Asheville, North Carolina
  - Novant Health Cancer Specialists, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Southern Oncology Specialists, Charlotte, North Carolina
  - Lake Norman Hematology Oncology Specialists, Huntersville, North Carolina
  - Novant Health Huntersville Medical Center, Huntersville, North Carolina
  - Southern Oncology Specialists, Huntersville, North Carolina
  - Novant Health Cancer Specialists, Matthews, North Carolina
  - Novant Health Matthews Medical Center, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists, Mooresville, North Carolina
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, William M. Cooper Pavilion, Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology PLLC, Gallatin, Tennessee
  - The West Clinic, P.C. d/b/a West Cancer Center, Germantown, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - The West Clinic, P.C. d/b/a West Cancer Center, Memphis, Tennessee
  - Tennessee Oncology PLLC, Murfreesboro, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Tennessee Oncology PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Shelbyville, Tennessee
  - Tennessee Oncology PLLC, Smyrna, Tennessee
  - The Center for Cancer and Blood Disorders, Arlington, Texas
  - Texas Oncology-South Austin, Austin, Texas
  - The Center for Cancer and Blood Disorders (Huguley), Burleson, Texas
  - Texas Oncology - Cedar Park, Cedar Park, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology-El Paso Cancer Treatment Center Grandview, El Paso, Texas
  - Texas Oncology-El Paso Cancer Treatment Center Gateway, El Paso, Texas
  - Texas Oncology - El Paso Cancer Treatment Center Joe Battle, El Paso, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Investigational Products Center (IPC), Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University Of Texas, Md Anderson Cancer Center, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center(IPC), Irving, Texas
  - Texas Oncology-Plano East, Plano, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Texas Oncology-Waco, Waco, Texas
  - The Center for Cancer and Blood Disorders, Weatherford, Texas
  - Virginia Cancer Specialists, PC, Alexandria, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
  - Northwest Cancer Specialists, P.C.(Admin Only), Vancouver, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- Australia (26):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - ICON Cancer Care (Haematology And Oncology Clinics Of Australasia (Hoca))-Milton, Milton, Queensland
  - Icon Cancer Care, Corporate Office, South Brisbane, Queensland
  - ICON Cancer Care, South Brisbane, Queensland
  - ICON Cancer Foundation, South Brisbane, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Adelaide Cancer Centre, Kurralta Park, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Cancer Care SA PTY Ltd, Kurralta Park, South Australia
  - Cancer Care SA trading as Icon Pharmacy Adelaide, Kurralta Park, South Australia
  - Victoria Breast and Oncology Care, East Melbourne, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Austin Health, Heidelberg Repatriation Hospital (radiology (MUGA)scans only), Heidelberg West, Victoria
  - Austin Health, The Austin Hospital, Melbourne, Victoria
  - Slade Pharmacy Mount Waverley, Mount Waverley, Victoria
  - Nova Pharmacy, Wendouree, Victoria
  - Ballarat Oncology & Haematology Services Clinical Trials Unit, Wendouree, Victoria
  - Ballarat Oncology & Haematology Services, Wendouree, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Sir Charles Gairdner Hospital Lung Institute Of Western Australia, Nedlands, Western Australia
  - River City Pharmacy, Auchenflower
  - Icon Cancer Care, Milton
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - CHU Sart Tilman Liege, Liège
- Brazil (13):
  - Instituto Nacional do Cancer Jose de Alencar Gomes da Silva, Rio de Janeiro, Rio de Janeiro
  - Central de Quimioterapia Hospital do Cancer-INCA-HCIII, Rio de Janeiro, Rio de Janeiro
  - Hospital do Cancer III - INCA / Instituto Nacional do Cancer / MS INCA HCIII, Rio de Janeiro, Rio de Janeiro
  - Hopital da Cidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital da Cidade de Passo Fundo - HCPF, Passo Fundo, Rio Grande do Sul
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao E Assistencia, Porto Alegre, Rio Grande do Sul
  - Hospital do Cancer de Barretos - Fundacao Pio XII, Barretos, São Paulo
  - Fundacao Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto de Oncologia de Piracicaba S/S Ltda., Piracicaba, São Paulo
  - Centro de Referencia da Saude da Mulher - Hospital Perola Byington, São Paulo, São Paulo
  - Clinica de Pesquisas e Centro de Estudos em Oncologia Ginecologica e Mamária Ltda., São Paulo, São Paulo
- France (11):
  - CHRU Jean Minjoz, Besançon
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Prive du Confluent, Nantes BP 20215
  - Hopital Saint Louis, Paris
  - Hopital Tenon, Paris
  - Institut de Cancerologie de l'Ouest - Site Rene Gauducheau, Saint-Herblain
  - Hopitaux Universitaires de Strasbourg - Hopital Civil, Strasbourg
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - CHU Bretonneau Centre Henry Kaplan, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (15):
  - Medizinisches Zentrum fur Hamatologie und Onkologie Munchen MVZ, Munich, Bavaria
  - Radiologicum, Munich, Bavaria
  - IOZ Muenchen, Munich, Bavaria
  - University of Munich (LMU), Grosshadern Hospital, Munich, Bavaria
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden, Dresden, Saxony
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Praxisklinik Krebsheilkunde fuer Frauen/Brustzentrum, Berlin
  - University Hospital Duesseldorf, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Klinik für Senologie / Brustzentrum, Essen
  - Universitaetsklinikum Freiburg, Klinik fuer Frauenheilunde, Freiburg im Breisgau
  - Oncologie Unter Ems, Leer
  - Klinikum rechts der Isar, TUM, Frauenklinik und Poliklinik, Munich
  - Unifrauenklinik am Klinikum Suedstadt, Rostock
  - Universitaetsfrauenklinik, Ulm
- Ireland (3):
  - Mater Misericordiae University Hospital, Dublin
  - St. Vincent's University Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (8):
  - Soroka University Medical Center, Beersheba
  - Oncology Institute, Rambam Health Care Campus, Haifa
  - Oncology Institute, Davidoff Center, Rabin Medical Center, Beilinson Campus, Petah Tikva
  - Division of Oncology Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Center, Tel Aviv
  - Oncology Institute, Assuta Medical Center, Tel Aviv
  - The Chaim sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin
- Italy (11):
  - A.O.S.G. Moscati - Contrada Amoretta, Avellino, AV
  - Ospedale S. Raffaelle di Milano, Milan, MI
  - A.S.S.T. Monza, Monza, Monza and Brianza
  - A.S.S.T. Monza, Oncologia Medica, Ospedale San Gerardo, Monza, Monza Brianza
  - La Maddalena Clinic For Cancer University Of Palermo, Palermo, PA
  - A.O.U. Pisana, DAI Oncologia, U.O. Oncologia Med. 2 Univ., Pisa, PI
  - Ospendale Sant'Andrea, Roma, RM
  - Ospedale Mater Salutis, Legnago, VR
  - S.S.D. Oncologia Medica Addarii - A.O.U. di Bologna - Policlinico Sant'Orsola-Malpighi, Bologna
  - Senologia Medica, IRCCS-Instituto Oncologico Europeo (IEO), Milan
  - Universita Campus Bio-Medico di Roma, Dipartimento Oncologia Medica, Roma
- Poland (19):
  - Centrum Terapii Wspolczesnej J.M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, LODZ Province
  - NZOZ Innowacyjna Medycyna, Dobra
  - Uniwersyteckie Centrum Kliniczne, Zaklad Medycyny Nuklearnej, Gdansk
  - Uniwersyteckie Centrum Kliniczne Klinika Onkologii i Radioterapii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Klinika Onkologii i Radioterapii, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Zaklad Radiologii, Gdansk
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Oddzial w Gliwicach, Gliwice
  - NU-MED Centrum Diagnostyki i Terapii Onkologicznej Katowice, Katowice
  - Uniwersyteckie Centrum Kliniczne im. Prof. K. Gibinskiego Slaskiego Uniwersytetu, Katowice
  - Europejskie Centrum Zdrowia Otwock Szpital im.F.Chopina, Otwock
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego, Poznan
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Pozna, Poznan
  - Szpital Kliniczny Przemienienia Panskiego Uniwersytetu Medycznego im. Karola, Poznan
  - Wielkopolskie Centrum Onkologii im. Marii Sklodowskiej-Curie, Poznan
  - Oddzial Onkologii Klinicznej, Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
  - Pracownia Tomografii Komputerowej , Samodzielny Publiczny Szpital Kliniczny Nr 2 PUM w Szczecinie, Szczecin
  - Pracownia Medycyny Nuklearnej, 109 Szpital Wojskowy z Przychodnia SP ZOZ, Szczecin
  - Centrum Onkologii - Instytut im. Marii Sklodowskiej-Curie Klinika Nowotworow Piersi i, Warsaw
  - Klinika Onkologii, Wojskowy lnstytut Medyczny, Warsaw
- Russia (3):
  - Gbuz Lood, Leningrad, Leningradskaya Oblast'
  - State Budgetary Institution of Healthcare "Republican Oncology dispensary"', Petrozavodsk
  - City Clinical Oncology Dispensary, Saint Petersburg
- South Korea (13):
  - Seoul National University Bundang Hospital, Bundang-gu, Gyeonggi-do
  - National Cancer Centre, Goyang-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Kyungpook National University Chilgok Hospital, Daegu
  - Gachon University Gil Medical Center, Incheon
  - Korea University Anam Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (17):
  - Centro Oncologico de Galicia, A Coruña
  - Hospital Nuestra Senora de Sonsoles(Complejo Asistencial de Avila), Ávila
  - Hospital Universitari Germans Trias i Pujol, Badalona Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic I Provincial, Barcelona
  - Consorcio Hospitalario Provincial de Castellon, Castellon
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitario de Canarias, La Laguna Santa Cruz de Tenerife
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Quiron Madrid, Pozuelo de Alarcon (Madrid)
  - Corporacio Sanitaria Parc Tauli, Sabadell Barcelona
  - Hospital Universitario Virgen Macarena, Seville
- Taiwan (4):
  - Changhua Christian Hospital, Changhua
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
- Ukraine (2):
  - Communal Institution "Krivorizhskiy Oncology Dispensary" of Dnipropetrovsk Regional Council, Kryvyi Rih
  - Regional Municipal Institution "Sumy Regional Clinical Oncology Dispensary", Thoracic Department, Sumy
- United Kingdom (6):
  - Sarah Cannon Research Institute UK, London, England
  - Nottingham University Hospital NHS Trust, Nottingham, Nottinghamshire
  - Royal Sussex County Hospital, Royal Alexandra Children's Hospital L10, Brighton
  - St James University Hospital, Leeds
  - Impretial College Healthcare NHS Trust, London
  - Cancer Research UK, Department of Medical Oncology - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Blum JL, Laird AD, Litton JK, Rugo HS, Ettl J, Hurvitz SA, Martin M, Roche HH, Lee KH, Goodwin A, Chen Y, Lanzalone S, Chelliserry J, Czibere A, Hopkins JF, Albacker LA, Mina LA. Determinants of Response to Talazoparib in Patients with HER2-Negative, Germline BRCA1/2-Mutated Breast Cancer. Clin Cancer Res. 2022 Apr 1;28(7):1383-1390. doi: 10.1158/1078-0432.CCR-21-2080. PMID 35091441
- [Derived] Ettl J, Quek RGW, Lee KH, Rugo HS, Hurvitz S, Goncalves A, Fehrenbacher L, Yerushalmi R, Mina LA, Martin M, Roche H, Im YH, Markova D, Bhattacharyya H, Hannah AL, Eiermann W, Blum JL, Litton JK. Quality of life with talazoparib versus physician's choice of chemotherapy in patients with advanced breast cancer and germline BRCA1/2 mutation: patient-reported outcomes from the EMBRACA phase III trial. Ann Oncol. 2018 Sep 1;29(9):1939-1947. doi: 10.1093/annonc/mdy257. PMID 30124753
- [Derived] Litton JK, Rugo HS, Ettl J, Hurvitz SA, Goncalves A, Lee KH, Fehrenbacher L, Yerushalmi R, Mina LA, Martin M, Roche H, Im YH, Quek RGW, Markova D, Tudor IC, Hannah AL, Eiermann W, Blum JL. Talazoparib in Patients with Advanced Breast Cancer and a Germline BRCA Mutation. N Engl J Med. 2018 Aug 23;379(8):753-763. doi: 10.1056/NEJMoa1802905. Epub 2018 Aug 15. PMID 30110579

RESULTS

PARTICIPANT FLOW:
Groups:
- Talazoparib: Participants received talazoparib 1 milligram (mg), orally, once daily until radiographic disease progression as determined by the central independent radiology facility (IRF), unacceptable toxicity, consent withdrawal, physician's decision to terminate treatment, or sponsor's decision to terminate the trial (up to a maximum of 70.2 months). One cycle was of 21 days.
- Physician's Choice Treatment: Participants received 1 of the following drugs in specified regimens, as per the physician's choice: 1) capecitabine 1250 milligram per meter square (mg/m^2) orally twice daily on Day 1 to 14 in each cycle; 2) eribulin mesylate 1.4 mg/m^2 (equivalent to eribulin 1.23 mg/ m^2), as 2 to 5 minute intravenous (IV) infusion on Day 1 and 8 in each cycle; 3) gemcitabine 1250 mg/m^2 as 30-minute IV infusion on Day 1 and 8 in each cycle; 4) vinorelbine 30 mg/m^2 as 6 to 10 minute IV infusion on Day 1, 8, and 15 in each cycle; until radiographic disease progression as determined by the central IRF, unacceptable toxicity, consent withdrawal, physician's decision to terminate treatment, or Sponsor's decision to terminate the trial (up to a maximum of 45.3 months). One cycle was of 21 days.
Period: Overall Study
Arm/Group | Talazoparib | Physician's Choice Treatment
Started | 287 | 144
Treated | 286 | 126
Completed | 0 | 0
Not Completed | 287 | 144
Not completed — Death | 214 | 98
Not completed — Lost to Follow-up | 12 | 7
Not completed — Withdrawal by Subject | 11 | 21
Not completed — Other | 50 | 18

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included all randomized participants.
Groups:
- Talazoparib: Participants received talazoparib 1 mg, orally, once daily until radiographic disease progression as determined by the central IRF, unacceptable toxicity, consent withdrawal, physician's decision to terminate treatment, or sponsor's decision to terminate the trial (up to a maximum of 70.2 months). One cycle was of 21 days.
- Physician's Choice Treatment: Participants received 1 of the following drugs in specified regimens, as per the physician's choice: 1) capecitabine 1250 mg/m^2 orally twice daily on Day 1 to 14 in each cycle; 2) eribulin mesylate 1.4 mg/m^2 (equivalent to eribulin 1.23 mg/ m^2), as 2 to 5 minute IV infusion on Day 1 and 8 in each cycle; 3) gemcitabine 1250 mg/m^2 as 30-minute IV infusion on Day 1 and 8 in each cycle; 4) vinorelbine 30 mg/m^2 as 6 to 10 minute IV infusion on Day 1, 8, and 15 in each cycle; until radiographic disease progression as determined by the central IRF, unacceptable toxicity, consent withdrawal, physician's decision to terminate treatment, or Sponsor's decision to terminate the trial (up to a maximum of 45.3 months). One cycle was of 21 days.
- Total: Total of all reporting groups
Arm/Group | Talazoparib | Physician's Choice Treatment | Total
Number analyzed (Participants) | 287 | 144 | 431
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (11.61) | 49.4 (12.12) | 48.1 (11.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 283 | 141 | 424
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 15 | 46
  Not Hispanic or Latino | 207 | 111 | 318
  Unknown or Not Reported | 49 | 18 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 31 | 16 | 47
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 1 | 12
  White | 190 | 108 | 298
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 55 | 19 | 74

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS): Independent Radiological Facility (IRF) Assessment
Description: IRF assessed PFS was defined as time (in months) from randomization until the date of first documented radiologic progressive disease per response evaluation criteria in solid tumors (RECIST) version 1.1 or death from any cause, whichever occurs first. As per RECIST v1.1, progression defined as 1) for target lesions: at least a 20% increase in the sum of target lesion measurements, compared to the smallest sum on study (including baseline), the absolute increase in the sum has to be at least 5 millimeter (mm); 2) for non-target lesions: unequivocal progression of non-target lesions, evaluated as a whole, such that it is clear that treatment has failed and disease is progressing, regardless of the status of the target lesions; 3) and/or appearance of one or more new lesions. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until radiologic progressive disease or death due to any cause (up to maximum duration of 36.9 months)
Population: Intent-to-treat (ITT) analysis population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 287 | 144
months | 8.6 [7.2 to 9.3] | 5.6 [4.2 to 6.7]
Statistical Analysis 1: Comparison: Talazoparib vs Physician's Choice Treatment; Hazard ratio was based on stratified Cox regression model with treatment as the only covariate (stratification factors: number of prior cytotoxic chemotherapy regimens, triple negative status, history of central nervous system metastasis status); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio, log = 0.542, 95% CI 2-sided [0.413 to 0.711]

2. Secondary Outcome: Percentage of Participants With Objective Response: Investigator Assessment
Description: Investigator assessed objective response was defined as the percentage of participants with a partial response (PR) or complete response (CR) as defined by RECIST v1.1. For target lesions: 1) CR: disappearance of all non-nodal target lesions. Target lymph nodes must reduce to less than 10 mm in short axis. 2) PR: At least a 30% decrease in the sum of diameters of target lesions, compared to the sum at baseline. For non-target lesions, CR: disappearance of all non-target lesions. Percentage of participants with objective response reported are based upon unconfirmed CR/PR.
Time Frame: Baseline until radiologic progressive disease or death due to any cause (up to a maximum duration of 36.9 months)
Population: ITT with measurable disease analysis population included all participants in the ITT population who had at least 1 target lesion identified at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 219 | 114
percentage of participants | 62.6 [55.78 to 68.99] | 27.2 [19.28 to 36.33]
Statistical Analysis 1: Comparison: Talazoparib vs Physician's Choice Treatment; p-value was based on stratified Cochran-Mantel-Haenszel method. Stratification factors: number of prior cytotoxic chemotherapy regimens, triple negative status, history of central nervous system metastasis status; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.99, 95% CI 2-sided [2.93 to 8.83]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in months) from randomization to death due to any cause. If death was not observed at the time of study cut-off date or permanently lost to follow-up, OS was censored at the date the participant was last known to be alive on or before the study cut-off date, whichever was earlier. The analysis was performed by Kaplan-Meier method.
Time Frame: Baseline until death due to any cause or analysis cut-off, up to a maximum duration of 61.4 months
Population: ITT analysis population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 287 | 144
months | 19.3 [16.6 to 22.5] | 19.5 [17.4 to 22.4]
Statistical Analysis 1: Comparison: Talazoparib vs Physician's Choice Treatment; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1693, Log Rank; Hazard Ratio (HR) = 0.848, 95% CI 2-sided [0.670 to 1.073]

4. Secondary Outcome: Trough Plasma Talazoparib Concentrations
Description: A predose PK sample was considered dose-compliant based on the following criteria: A participant must have received 21 consecutive days of 1 mg talazoparib without dosing interruption prior to sample collection; and the predose PK sample must have been collected 24 hours +/- 10 percent (2 hours and 24 minutes) after the previous day's dose and no more than 5 minutes (0.083 hours) after the administration of the dose on the day of PK sample collection.
Time Frame: Predose on Day 1 of Cycle 2, 3 and 4
Population: Analysis population included participants who received at least 1 dose of talazoparib and had dose compliant pharmacokinetic (PK) predose sample. Here, "number analyzed" signifies number of participants who were evaluable for the specified categories. This endpoint was not planned to be analyzed for the reporting arm "Physician's Choice Treatment".
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picogram per milliliter (pg/mL)
Arm/Group | Talazoparib
Number analyzed (Participants) | 175
Picogram per milliliter (pg/mL)
  Cycle 2 Day 1: Predose: number analyzed (Participants) | 137
  Cycle 2 Day 1: Predose | 3370 (76.9)
  Cycle 3 Day 1: Predose: number analyzed (Participants) | 120
  Cycle 3 Day 1: Predose | 3570 (49.9)
  Cycle 4 Day 1: Predose: number analyzed (Participants) | 107
  Cycle 4 Day 1: Predose | 3400 (48.4)

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse events (AE) was any untoward medical occurrence (e.g., sign, symptom, illness, disease or injury) in a participant administered study drug or other protocol-imposed intervention, regardless of attribution. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug or the day before initiation of a new antineoplastic therapy or 30 days after the date of the last dose date of study drug, whichever occurred first, that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and all non-SAEs.
Time Frame: Talazoparib: Baseline up to a maximum duration of 71.3 months; Physician's Choice Treatment: Baseline up to maximum duration of 46.1 months
Population: Safety analysis population included all participants who received at least 1 dose of any study drug (talazoparib or protocol-specified PCT).
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 286 | 126
Participants
  TEAEs | 282 | 123
  SAEs | 103 | 39

6. Secondary Outcome: Number of Participants With Grade 3 or 4 Post-baseline Toxicities in Laboratory Parameters: Hematology
Description: Toxicity grades were evaluated based on as National Cancer Institute Common Toxicity Criteria for Adverse Events Version 4.03 (NCI CTCAE v4.03). NCI CTCAE v4.03 defined the severity grade as: grade 1 (mild), grade 2 (moderate), grade 3 (severe), grade 4 (potentially life threatening) and grade 5 (death related to AE) for each parameter. Key hematology parameters included hemoglobin (gram per liter [g/L]), leukocytes (10^6 cells per liter), lymphocytes (10^6 cells per liter), neutrophils (10^6 cells per liter), and platelets (10^9 cells per liter). Low value indicated lower values than the baseline values and high value indicated higher values than the baseline values. Only those categories in which at least 1 participant had data were reported.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 286 | 126
Participants
  Hemoglobin: Low value | 115 | 8
  Leukocytes: Low value | 43 | 31
  Lymphocytes: Low value | 54 | 11
  Neutrophils: Low value | 65 | 48
  Platelets: Low value | 44 | 2

7. Secondary Outcome: Number of Participants With Grade 3 or 4 Post-baseline Toxicities in Laboratory Parameters: Chemistry
Description: Toxicity grades were evaluated based on as NCI CTCAE v4.03. NCI CTCAE v4.03 defined the severity grade as: grade 1 (mild), grade 2 (moderate), grade 3 (severe) and grade 4 (potentially life threatening) and grade 5 (death related to AE) for each parameter. Key chemistry parameters included alanine aminotransferase (units per liter), alkaline phosphatase (units per liter), aspartate aminotransferase (units per liter) and bilirubin (micromole per liter). High value indicated higher values than the baseline values and low value indicated lower values than the baseline values. Only those categories in which at least 1 participant had data were reported.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 286 | 126
Participants
  Alanine Aminotransferase: High Value | 5 | 3
  Alkaline Phosphatase: High Value | 6 | 2
  Aspartate Aminotransferase: High Value | 7 | 4
  Bilirubin: High Value | 4 | 1

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Changes From Baseline in Vital Signs
Description: Criteria for potentially clinically significant changes in vital signs included a) Systolic blood pressure: 1) absolute results (AB) greater than (>) 180 millimeter of mercury (mmHg) and increase from baseline (IFB) greater than or equal to (>=) 40 mmHg, 2) absolute results less than (<) 90 mmHg and decrease from baseline (DFB) >30 mmHg; b) Diastolic blood pressure: 1) absolute results >110 mmHg and >=30 mmHg increase from baseline, 2) absolute results <50 mmHg and >20 mmHg decrease from baseline 3) >=20 mmHg increase from baseline; c) Heart rate: 1) absolute results>120 beats per minute [bpm] and >30 bpm increase from baseline, 2) absolute results <50 bpm and >20 bpm decrease from baseline and d) Weight: >10 percent [%] decrease from baseline.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 286 | 126
Participants
  SBP: AB>180 mmHg and IFB >=40 mmHg | 3 | 2
  SBP: AB<90 mmHg and DFB >30 mmHg | 8 | 2
  DBP: AB>110 mmHg and IFB >=30 mmHg | 0 | 0
  DBP: AB<50 mmHg and DFB>20 mmHg | 15 | 7
  DBP: IFB>=20 mmHg | 39 | 13
  Heart rate: AB >120 bpm and IFB >30 bpm | 6 | 2
  Heart rate: AB <50 bpm and DFB >20 bpm | 2 | 0
  Weight: >10% DFB | 23 | 13

9. Secondary Outcome: Number of Participants Taking At-least One Concomitant Medication
Description: Any medication (other than study drug) which was administered to participants during study after first dose of study drug were considered as concomitant medications.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 286 | 126
Participants | 281 | 126

10. Other Pre Specified Outcome: Duration of Response (DOR): Investigator Assessment
Description: DOR = time from first radiographic documentation of OR (PR or CR) till radiographic disease progression (PD) as per RECIST v1.1 by investigator assessment or to death due to any cause, whichever was first. RECIST 1.1, a) target lesion (TL): CR= disappearance of all non-nodal TL, target lymph nodes reduce to <10 mm in short axis, PR= at least 30% decrease in sum of diameters of TL, compared to the sum at baseline, PD= at least 20% increase in sum of TL measurements, compared to smallest sum on study including baseline, absolute increase in sum has to be at least 5 mm; b) for non-TL: CR= disappearance of all non-TL, PD= unequivocal progression of non-TL, such that treatment has failed, disease is progressing, regardless of status of TL; c) PD =and/or appearance of >=1 new lesions. DOR = (earliest date of progression, death, or censoring-date of first documented OR + 1)/30.4375. Analysis was performed by Kaplan-Meier method.
Time Frame: From first documentation of CR or PR until disease progression or death due to any cause, whichever occurred first (up to 36.9 months)
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 219 | 114
months | 5.4 [2.8 to 11.2] | 3.1 [2.4 to 6.7]

11. Other Pre Specified Outcome: Change From Baseline in Global Health Status/Quality of Life (QoL) Measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) at Average Duration Over Week 4 up to Week 160
Description: EORTC QLQ-C30: cancer-specific instrument with 30 questions to assess the participant QoL. First 28 questions used to evaluate 5 functional scales (physical, role, cognitive, emotional, social), 3 symptom scales (fatigue, nausea and vomiting, pain) and other single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, financial difficulties). Each question assessed on 4-point scale (1= not at all, 2= a little, 3= quite a bit, 4= very much); functional scales: higher score = better level of functioning; symptom scale: higher score = more severe symptoms; for single items: higher score= more severe problem. Last 2 questions used to evaluate global health status (GHS)/QoL. Each question was assessed on 7-point scale (1= very poor to 7= excellent). Scores averaged, transformed to 0-100 scale; higher score=better quality of life/better level of functioning. Change from baseline was calculated by subtracting the baseline value from the average value of Week 4 to 160.
Time Frame: Baseline, Week 4 up to Week 160
Population: Patient-reported outcomes (PRO) evaluable population included all participants who completed the PRO questionnaire at baseline and at least 1 visit post-baseline.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 262 | 114
units on a scale | 3.0 [1.2 to 4.8] | -5.4 [-8.8 to -2.0]
Statistical Analysis 1: Comparison: Talazoparib vs Physician's Choice Treatment; Analysis was based on repeated measures mixed-effect model with an intercept term, treatment, time, treatment-by-time, and baseline as covariate. Analysis was based on restricted maximum likelihood using unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 8.4, 95% CI 2-sided [4.6 to 12.3]

12. Other Pre Specified Outcome: Time to Deterioration (TTD) in Global Health Status/Quality of Life (QOL)
Description: TTD in global health status (GHS)/QoL=time (in months) from randomization to the first observation with >=10 point decrease and no subsequent observations with<10 point decrease from baseline in GHS/QoL score based on EORTC-QLQ-C30. EORTC QLQ-C30 is a cancer-specific instrument with 30 questions to assess participant quality of life. Question 29 and 30 were used to evaluate GHS/QoL. Each question was assessed on a 7-point scale (1=very poor to 7=excellent). Scores averaged, transformed to 0-100 scale; higher score=better quality of life/better level of functioning.
Time Frame: Baseline up to a maximum duration of 36.9 months
Population: PRO-evaluable population included all participants who completed the PRO questionnaire at baseline and at least 1 visit post-baseline.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 262 | 114
months | 24.3 [13.8 to NA] — Upper limit of 95% CI was not estimable, since only few participants had event. | 6.3 [4.9 to 12.2]
Statistical Analysis 1: Comparison: Talazoparib vs Physician's Choice Treatment; Hazard ratio is based on stratified Cox regression model with treatment as the only covariate (stratification factors: number of prior cytotoxic chemotherapy regimens, triple negative status, history of central nervous system metastasis status); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.376, 95% CI 2-sided [0.257 to 0.549]

13. Other Pre Specified Outcome: Time to Deterioration (TTD) in Breast Symptoms Scale as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Breast Cancer Module (EORTC-QLQ-BR23)
Description: TTD was defined as the time (in months) from randomization to the first observation with a>=10 point increase and no subsequent observations with a <10 point increase from baseline in breast symptom score based on the EORTC-QLQ-BR23. EORTC-QLQ-BR23 is a disease-specific module for breast cancer developed as a supplement for the EORTC-QLQ-C30 to assess the quality of life of participants with breast cancer. EORTC-QLQ-BR23 symptoms subscale includes 4 items: systemic therapy side effects, breast symptoms, arm symptoms, upset by hair loss. Each item is rated by choosing 1 of 4 possible responses that record the level of intensity (1= not at all, 2= a little, 3= quite a bit, and 4= very much), higher scores=high level of symptom/problems.
Time Frame: Baseline up to a maximum duration of 36.9 months
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Talazoparib | Physician's Choice Treatment
Number analyzed (Participants) | 262 | 114
months | NA [NA to NA] — Median and 95% CI was not estimable due to the low number of participants with event. | NA [10.3 to NA] — Median and upper limit of 95% CI was not estimable due to the low number of participants with event.
Statistical Analysis 1: Comparison: Talazoparib vs Physician's Choice Treatment; Hazard ratio is based on stratified Cox regression model with treatment as the only covariate (stratification factors: number of prior cytotoxic chemotherapy regimens, triple negative status, history of central nervous system); Test type: Superiority; p = 0.0053, Log Rank; Hazard Ratio (HR) = 0.392, 95% CI 2-sided [0.198 to 0.775]

ADVERSE EVENTS:
Time Frame: Talazoparib: Baseline up to a maximum duration of 71.3 months; Physician's Choice Treatment: Baseline up to maximum duration of 46.1 months
Description: Same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AEs and SAEs were collected for safety population.
Arm/Group | Talazoparib | Physician's Choice Treatment
All-Cause Mortality (participants affected / at risk) | 220/286 | 100/126
Serious Adverse Events (participants affected / at risk) | 103/286 | 39/126
Other Adverse Events (participants affected / at risk) | 282/286 | 123/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib (N=286) | Physician's Choice Treatment (N=126)
Anaemia (Blood and lymphatic system disorders) | 18 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 3 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Diplopia (Eye disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 8 | 2
General physical health deterioration (General disorders) | 2 | 2
Non-cardiac chest pain (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Discomfort (General disorders) | 0 | 1
Localised oedema (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 0 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 2
Cytomegalovirus infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Anal abscess (Infections and infestations) | 1 | 0
Breast cellulitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Scar (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 4 | 0
Neutrophil count decreased (Investigations) | 1 | 2
Hepatic enzyme increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 5 | 0
Seizure (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Bartholin's cyst (Reproductive system and breast disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0
Breast reconstruction (Surgical and medical procedures) | 1 | 0
Salpingo-oophorectomy (Surgical and medical procedures) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Lymphadenectomy (Surgical and medical procedures) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib (N=286) | Physician's Choice Treatment (N=126)
Anaemia (Blood and lymphatic system disorders) | 153 | 24
Neutropenia (Blood and lymphatic system disorders) | 77 | 36
Thrombocytopenia (Blood and lymphatic system disorders) | 50 | 7
Leukopenia (Blood and lymphatic system disorders) | 24 | 12
Lacrimation increased (Eye disorders) | 10 | 9
Nausea (Gastrointestinal disorders) | 142 | 60
Diarrhoea (Gastrointestinal disorders) | 68 | 32
Vomiting (Gastrointestinal disorders) | 74 | 28
Constipation (Gastrointestinal disorders) | 66 | 28
Abdominal pain (Gastrointestinal disorders) | 36 | 18
Dyspepsia (Gastrointestinal disorders) | 33 | 10
Stomatitis (Gastrointestinal disorders) | 24 | 7
Dry mouth (Gastrointestinal disorders) | 19 | 8
Fatigue (General disorders) | 147 | 54
Asthenia (General disorders) | 45 | 12
Pyrexia (General disorders) | 31 | 21
Oedema peripheral (General disorders) | 23 | 8
Mucosal inflammation (General disorders) | 16 | 9
Non-cardiac chest pain (General disorders) | 17 | 5
Influenza like illness (General disorders) | 20 | 2
Upper respiratory tract infection (Infections and infestations) | 41 | 13
Viral upper respiratory tract infection (Infections and infestations) | 35 | 8
Urinary tract infection (Infections and infestations) | 30 | 3
Sinusitis (Infections and infestations) | 21 | 4
Neutrophil count decreased (Investigations) | 30 | 18
Weight decreased (Investigations) | 23 | 15
Platelet count decreased (Investigations) | 36 | 4
White blood cell count decreased (Investigations) | 32 | 5
Aspartate aminotransferase increased (Investigations) | 15 | 15
Alanine aminotransferase increased (Investigations) | 11 | 15
Decreased appetite (Metabolism and nutrition disorders) | 62 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 67 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 55 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 45 | 14
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 28 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 25 | 14
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 29 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 17 | 6
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 7
Muscle spasms (Musculoskeletal and connective tissue disorders) | 18 | 3
Headache (Nervous system disorders) | 96 | 29
Dizziness (Nervous system disorders) | 51 | 13
Dysgeusia (Nervous system disorders) | 30 | 11
Paraesthesia (Nervous system disorders) | 13 | 15
Neuropathy peripheral (Nervous system disorders) | 19 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 7
Insomnia (Psychiatric disorders) | 38 | 10
Anxiety (Psychiatric disorders) | 24 | 9
Depression (Psychiatric disorders) | 24 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 65 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 78 | 35
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4 | 28
Rash (Skin and subcutaneous tissue disorders) | 29 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 14 | 9
Hot flush (Vascular disorders) | 23 | 9
Abdominal pain upper (Gastrointestinal disorders) | 28 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT01945775/Prot_001.pdf
  • Statistical Analysis Plan (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/75/NCT01945775/SAP_000.pdf